CLINICAL TRIAL: NCT02992197
Title: A Double-blind, Randomized Controlled Trial of the Effect of Vaccine Inoculum on Oral Rotavirus Vaccine (Rotarix, GlaxoSmithKline) Take and Immunogenicity in Dhaka, Bangladesh
Brief Title: The Effects of Increased Inoculum on Oral Rotavirus Vaccine Take and Immunogenicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Charles H. Hood Foundation (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Benjamin Lee, Assistant Professor, Department of Pediatrics, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHRMS 17-0166
Record Dates: First submitted 2016-12-01; First posted 2016-12-14 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Rotavirus Infection; Vaccine Response Impaired; Vaccine Virus Shedding
Keywords: Rotavirus; Oral vaccines; Vaccine underperformance; Vaccine shedding
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotarix, single dose (Active Comparator): Rotarix 1.5 mL (standard single dose) and 1.5 mL of placebo by mouth (sterile, pharmacy-grade water) at both 6 and 10 weeks of life
  Interventions: Biological: Rotarix, dose 1; Drug: Placebo (for Rotarix dose 2)
- Rotarix, double dose (Experimental): Rotarix 3 mL by mouth (two standard doses administered simultaneously) at both 6 and 10 weeks of life
  Interventions: Biological: Rotarix, dose 1; Biological: Rotarix, dose 2

INTERVENTIONS:
Biological: Rotarix, dose 1 — Rotarix, dose 1
Biological: Rotarix, dose 2 — Rotarix, dose 2
  Arms: Rotarix, double dose
Drug: Placebo (for Rotarix dose 2) — Sterile water to provide volume equivalent as a second dose of Rotarix
  Arms: Rotarix, single dose

SUMMARY:
Rotavirus is the leading cause of diarrhea in children worldwide. Oral rotavirus vaccines work remarkably well in high-income countries, but for unclear reasons they underperform in low-income countries. A double-blind, randomized control trial will be performed to evaluate whether using a higher dose of a currently licensed vaccine (Rotarix, GlaxoSmithKline) can improve immune responses among infants in Dhaka, Bangladesh.

Infants will be randomized 1:1 to receive either a standard or a double dose of Rotarix at 6 and 10 weeks of life. Infants will be assessed for fecal vaccine shedding and serum rotavirus-specific IgA responses to determine vaccine immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy infant (as determined by medical officers)
2. Age 0-7 days at enrolment
3. Mother willing and able to provide signed informed consent
4. Mother willing to allow infant to be vaccinated according to study schedule
5. Mother willing to allow biological specimens, including blood, stool, and saliva, to be collected from infant according to study protocol
6. Mother willing and able to adhere to study schedule

Exclusion Criteria:

1. Obvious congenital malformation
2. Birth weight (if known) or enrolment weight (if birth weight unknown) < 2000 gm
3. Known immunocompromising condition in infant
4. Enrolment in other vaccine research trials
5. Other household member enrolled in this study

Max Age: 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lee, M.D., Principal Investigator — University of Vermont
Locations (1):
- International Center for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee B, Dickson DM, Alam M, Afreen S, Kader A, Afrin F, Ferdousi T, Damon CF, Gullickson SK, McNeal MM, Bak DM, Tolba M, Carmolli MP, Taniuchi M, Haque R, Kirkpatrick BD. The effect of increased inoculum on oral rotavirus vaccine take among infants in Dhaka, Bangladesh: A double-blind, parallel group, randomized, controlled trial. Vaccine. 2020 Jan 3;38(1):90-99. doi: 10.1016/j.vaccine.2019.09.088. Epub 2019 Oct 10. PMID 31607603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose
Started | 110 | 110
Completed | 99 | 103
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Population: The a priori primary analysis was designed to evaluate study outcomes among those who completed the study per-protocol. Due to anticipated levels of attrition, the per-protocol population differs from the total numbers of initial enrollees. Data presented are for the per protocol population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose | Total
Number analyzed (Participants) | 97 | 92 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 97 | 92 | 189
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 4.8 (1.8) | 5.0 (1.8) | 4.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 41 | 92
  Male | 46 | 51 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bangladesh | 97 | 92 | 189
Birth place [Count of Participants; unit: Participants]
  Home birth | 19 | 25 | 44
  Hospital/clinic birth | 78 | 67 | 145
Mode of delivery [Count of Participants; unit: Participants]
  Vaginal | 55 | 50 | 105
  Caesarean section | 42 | 42 | 84
Weight [Mean (Standard Deviation); unit: kg] | 2.81 (0.44) | 2.86 (0.38) | 2.83 (0.42)
Length [Mean (Standard Deviation); unit: cm] | 48.9 (2.6) | 48.7 (0.21) | 48.8 (2.2)
Head circumference [Mean (Standard Deviation); unit: cm] | 34.1 (1.3) | 34.2 (1.3) | 34.1 (1.3)
Water treatment [Count of Participants; unit: Participants]
  None | 24 | 29 | 53
  Water filter | 4 | 2 | 6
  Boil | 69 | 61 | 130
Type of toilet [Count of Participants; unit: Participants]
  Septic tank or toilet | 52 | 45 | 97
  Water-sealed or slab latrine | 41 | 44 | 85
  Pit latrine or open latrine | 4 | 3 | 7
  Open drain beside home | 44 | 55 | 99
Family demographics [Count of Participants; unit: Participants]
  Mother's education <= secondary | 81 | 74 | 155
  Father's education <= secondary | 71 | 72 | 143
  Homeowner | 43 | 32 | 75
  Any food deficit | 31 | 37 | 68
  Municipal (piped) water source | 93 | 80 | 173
Monthly household income in Taka [Median (Inter-Quartile Range); unit: Taka] | 15000 [10000 to 20000] | 15000 [10000 to 20000] | 15000 [10000 to 20000]

OUTCOME MEASURES:

1. Primary Outcome: Number (or Percentage) of Infants in Each Study Arm Who Test Positive for Fecal Rotavirus Vaccine-strain Virus Shedding Post-vaccination
Description: This will be an aggregate measure demonstrating a change from baseline. Infants will have stool collected immediately prior to Rotarix vaccination at weeks 6 and 10 of life, then 4, 7, and 14 days following each dose (i.e. last assessment at week 12 of life). Each specimen will be assessed for vaccine-strain virus (i.e. fecal vaccine shedding) at each time point by polymerase chain reaction. Any child who has a change in fecal vaccine shedding status, from negative at baseline (6 weeks) to positive at any subsequent time point, will be categorized as having met the outcome measure for positive fecal vaccine shedding.
Time Frame: Measured through week 12 of life
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose
Number analyzed (Participants) | 97 | 92
Participants | 63 | 55

2. Primary Outcome: Number (or Percentage) of Infants in Each Study Arm With Rotavirus-specific Plasma Immunoglobulin A (IgA) Seroconversion Post-vaccination
Description: This outcome will measure seroconversion, i.e. the change in plasma rotavirus-specific IgA concentration at week 14 of life compared to week 6 of life (baseline). Blood will be collected from infants prior to the first dose of Rotarix at week 6 of life and again at week 14 of life (4 weeks following the second dose) for measurement of plasma rotavirus-specific IgA by enzyme immunoassay. Infants will be assessed for seroconversion (IgA concentration <=20 U/mL pre-vaccination and >20 post-vaccination). Infants who demonstrate rotavirus-specific IgA seroconversion will be categorized as having met the outcome measure.
Time Frame: Measured at week 14 of life
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose
Number analyzed (Participants) | 97 | 92
Participants | 41 | 42

3. Primary Outcome: Number (or Percentage) of Infants in Each Study Arm With Successful Vaccine Take, Defined as Positive Fecal Vaccine Shedding Post-vaccination OR Rotavirus-specific Plasma IgA Seroconversion Post-vaccination
Description: Vaccine take is an aggregate, dichotomous immunogenicity measure (successful vaccine take vs no vaccine take). Infants positive for either fecal vaccine shedding OR plasma rotavirus-specific IgA seroconversion (as described in Outcomes 1 and 2, respectively) will be categorized as having met the outcome measure of successful vaccine take. Those who met neither outcome will be categorized as no vaccine take.
Time Frame: Measured at week 14 of life
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose
Number analyzed (Participants) | 97 | 92
Participants | 69 | 62

ADVERSE EVENTS:
Time Frame: Enrollment (<7 days of life) through week 14 study visit (4 months) for serious adverse events; week 6 visit (first vaccine dose) through Week 14 visit + 3 days (end of participation) for all other AEs (2 months)
Description: Serious adverse events were recorded from study enrollment (<7 days of life) but all other adverse events were only recorded starting from the first study intervention (at the week 6 clinic visit), the total numbers of children evaluated for serious adverse events (which is based on study enrollment) differs from those evaluated for adverse events (which is based on the number of children dosed starting at week 6 of life, and is less due to attrition between enrollment and first dosing).
Arm/Group | Rotarix, Single Dose | Rotarix, Double Dose
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 2/110 | 4/110
Other Adverse Events (participants affected / at risk) | 28/107 | 31/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotarix, Single Dose (N=110) | Rotarix, Double Dose (N=110)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 2 (4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subacute intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotarix, Single Dose (N=107) | Rotarix, Double Dose (N=106)
Diarrhea (Gastrointestinal disorders) | 18 (20) | 16 (17)
Cough or runny nose (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 18 (19)
Gastroenteritis (vomiting and/or diarrhea) (Gastrointestinal disorders) | 19 (21) | 18 (21)
Respiratory tract infection (Infections and infestations) | 22 (24) | 21 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02992197/Prot_SAP_000.pdf